CLINICAL TRIAL: NCT02042274
Title: Omega-3 Fatty Acids and Genes Interact to Influence Cardiometabolic Health.
Brief Title: Efficacy Study Regarding the Beneficial Effects of Omega-3 Fatty Acids on Cardiometabolic Health
Acronym: FOHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, David M Mutch, Associate Professor, University of Guelph
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fish Oil and Health Study; 12JL006 (Other: University of Guelph)
Record Dates: First submitted 2014-01-20; First posted 2014-01-22 (Estimated); Results first posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-02

CONDITIONS: Metabolic Syndrome X
Keywords: Fish oil; EPA; DHA; fatty acids; genetic variation; gene expression
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fish oil supplement (Experimental): Fish oil supplements providing up to 3g per day of EPA and DHA
  Interventions: Dietary Supplement: Fish oil supplement

INTERVENTIONS:
Dietary Supplement: Fish oil supplement — Participants are instructed to consume fish oil supplements on a daily basis for a 3-month period.
  Other Names: Jamieson Omega-3 complete supplements; Ocean Nutrition MEG-3 supplements

SUMMARY:
Fish oil supplements (which are rich in omega-3 fatty acids) have been shown to provide cardiometabolic benefits to individuals of all ages. Specifically, the daily consumption of fish oil supplements has been reported to reduce blood triglyceride levels, and influence glucose homeostasis and whole-body inflammation. However, recent evidence highlights important gaps in our understanding with respect to the impact of fish oil supplements on health; specifically, not everyone responds to these supplements in the same manner. The goal of this research is to explore how an individual's genetic make-up may modify their response to fish oil supplements.

DETAILED DESCRIPTION:
The typical Western diet is now recognized to have insufficient amounts of omega-3 fatty acids (in particular EPA and DHA). These fatty acids have several known health benefits, including improvements in heart health, metabolic syndrome, and inflammation. These benefits occur because omega-3 fatty acids can regulate a myriad of cellular functions. In order to increase the levels of these omega-3 fatty acids in the body, individuals must either consume more marine products or take an omega-3 rich dietary supplement, such as fish oil. While fish oil supplements are commonly consumed by people, it is now recognized that not everyone responds to these supplements in the same manner. Therefore this study aims to improve our understanding of why people respond differently to the same dietary supplement. The goals of this research will be accomplished using a number of approaches:

1. The investigators will examine how fish oil supplementation leads to an enrichment of EPA and DHA in various cells throughout the body (erythrocytes, adipose tissue, etc).
2. The investigators will determine the dynamic changes in EPA and DHA incorporation into different cell-types during distinct phases of our dietary intervention study (e.g. during supplementation and subsequent wash out periods).
3. The investigators will study how fish oil supplements influence various blood markers of cardiometabolic health (e.g. triglycerides, cholesterol, glucose, C-reactive protein, etc) and whether this is modulated by an individual's genotype.

ELIGIBILITY:
Inclusion Criteria:

* between 18-25 years old
* male
* good general health

Exclusion Criteria:

* currently taking a fish oil supplement
* currently taking an omega-3 supplement
* currently consuming a diet high in omega-3 (high in ALA, EPA, or DHA)
* not able to maintain a consistent lifestyle routine throughout the study duration
* have an allergy which would prevent them from taking a fish oil pill
* schedule conflict with study visits
* overweight or obese

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Mutch, PhD, Principal Investigator — University of Guelph
Locations (1):
- University of Guelph - Human Nutraceutical Research Unit, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Roke K, Mutch DM. The role of FADS1/2 polymorphisms on cardiometabolic markers and fatty acid profiles in young adults consuming fish oil supplements. Nutrients. 2014 Jun 16;6(6):2290-304. doi: 10.3390/nu6062290. PMID 24936800

RESULTS

PARTICIPANT FLOW:
Groups:
- Fish Oil Supplement: Fish oil supplements providing up to 3g per day of EPA and DHA
  Fish oil supplement: Participants are instructed to consume fish oil supplements on a daily basis for a 3-month period.
  Measurements are made at three time points: Baseline (Day 0 - before beginning fish oil supplementation), 3 months (Day 90 - after fish oil supplementation), and 5 months (Day 150 - 2 month washout).
Period: Overall Study
Arm/Group | Fish Oil Supplement
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Fish Oil: Fish oil supplements providing up to 3g per day of EPA and DHA, for 90 days.
Arm/Group | Fish Oil
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Region of Enrollment [Count of Participants; unit: Participants] — Subjects were recruited through a poster campaign at the University of Guelph campus.
  Participants
    Canada | 12
Triglycerides [Mean (Standard Deviation); unit: mmol/L] | 0.9 (0.3)

OUTCOME MEASURES:

1. Primary Outcome: Blood Triglyceride
Description: Blood triglycerides were measured at distinct time points: baseline, after 3 months supplementation, and after a 2 month wash out period.
Time Frame: Baseline, 3 months, 5 months
Population: Healthy adults, ranging in age from 18-65 years.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Fish Oil Supplement
Number analyzed (Participants) | 12
mmol/L
  Baseline | 0.9 (0.3)
  3 Months | 0.8 (0.3)
  5 months | 0.9 (0.5)

2. Secondary Outcome: Blood Glucose
Description: Blood glucose levels measured at distinct time points: baseline, after 3 months supplementation, and after a 2 month wash out period.
Time Frame: Baseline, 3 months, 5 months
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Fish Oil Supplement
Number analyzed (Participants) | 12
mmol/L
  Baseline | 4.4 (1.4)
  3 Months | 3.9 (1.3)
  5 months | 4.2 (1.4)

ADVERSE EVENTS:
Time Frame: Through study completion (total of 5 months)
Arm/Group | Fish Oil Supplement
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No